CLINICAL TRIAL: NCT00657306
Title: Adrenal Insufficiency in Cirrhotics With Ascites. Effects of Stress Doses of Hydrocortisone on Renal Function and on Liver and Systemic Haemodynamics
Brief Title: Adrenal Insufficiency in Cirrhotics With Ascites. Effects of Hydrocortisone on Renal and Haemodynamic Function
Acronym: AILD
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Turin, Italy (Other)
Responsible Party: AOU San Giovanni Battista di Torino, Carlo Alessandria
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AILD
Record Dates: First submitted 2008-04-09; First posted 2008-04-14 (Estimated); Last update posted 2008-04-14 (Estimated); Status verified 2008-04

CONDITIONS: Cirrhosis With Ascites
Keywords: Cirrhosis; Ascites; Adrenal insufficiency; Hepatorenal syndrome; Portal hypertension
MeSH Terms: conditions — Fibrosis; Ascites; Adrenal Insufficiency; Hepatorenal Syndrome; Hypertension, Portal | interventions — Hydrocortisone

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Hydrocortisone, 50 mg/6 h per day
  Interventions: Drug: hydrocortisone
- 2 (Placebo Comparator): dextrose solution 5%
  Interventions: Drug: dextrose solution 5%

INTERVENTIONS:
Drug: hydrocortisone — 50 mg/6 h per day
  Arms: 1
Drug: dextrose solution 5% — dextrose solution 5% 100 ml/6 h per day
  Arms: 2

SUMMARY:
Relative adrenal insufficiency (RAI) is an well known condition in patients with septic shock. Liver failure (including chronic liver failure)and sepsis are both characterized by hyperdynamic circulatory failure (with low arterial pressure) and high levels of pro-inflammatory cytokines.

Hydrocortisone has been shown to have a beneficial effect on clinical outcome. The aim of this study is to evaluate the incidence of RAI in the different settings of ascites in cirrhosis and the usefulness of hydrocortisone in this context.

ELIGIBILITY:
Inclusion Criteria:

* Cirrhosis with ascites, with or without hepatorenal syndrome

Exclusion Criteria:

* Age < 18 and > 75 years
* Shock or bacterial infection present at the inclusion or during the previous week
* Bleeding present at the inclusion or during the previous week
* Multifocal HCC
* Organic renal failure
* Hearth or pulmonary failure

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2008-05; Primary Completion 2008-12 (Estimated); Study Completion 2009-05 (Estimated)

PRIMARY OUTCOMES:
renal function | 10 days

CONTACTS AND LOCATIONS:
Overall Officials: Carlo Alessandria, MD, Principal Investigator — Division of gastroenterology and hepatology
Locations (1):
- San Giovanni Battista Hospital, Turin, Italy